CLINICAL TRIAL: NCT04913467
Title: Potential Effects of Ileocolonic Delivered Vitamins or the Groningen Anti-Inflammatory Diet on Course of Crohn's Disease and the Microbiome of Healthy Volunteers: a Randomized Controlled Trial - The Vita-GrAID Study
Brief Title: Effect of Ileocolonic Delivered Vitamins and an Anti-Inflammatory Diet on Crohn's Disease and Healthy Volunteers
Acronym: Vita-GrAID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof. dr. G. Dijkstra, Clinical Professor, Head of Inflammatory Bowel Disease Center and Intestinal Transplantation Center, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL66008.056.20; 202000683 (Other: UMCG)
Record Dates: First submitted 2021-05-03; First posted 2021-06-04 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Crohn Disease
Keywords: Inflammatory Bowel Disease; IBD; Crohn; Vitamins; Diet; Riboflavin; Ascorbic Acid; Niacin; Microbiome
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, partly blinded, multicenter clinical food trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Groningen Anti-Inflammatory Diet (GrAID) (Experimental): Specially designed diet based on the most recent scientific evidence of the inflammatory characteristics of food and food groups.
  Interventions: Other: Groningen Anti-Inflammatory Diet (GrAID)
- ColoVit capsule (Experimental): 2 times daily intake of a supplement containing 37,5 mg vitamin B2, 2,5 mg vitamin B3 and 250 mg vitamin C in a ColoPulse-coated capsule, a pH-sensitive coating allowing ileocolonic-targeted-delivery
  Interventions: Dietary Supplement: ColoVit capsule
- Placebo capsule (Placebo Comparator): 2 times daily intake of a capsule containing microcrystalline cellulose which is coated using the same ColoPulse technology as is used with the ColoVit
  Interventions: Other: ColoPulse-placebo capsule

INTERVENTIONS:
Other: Groningen Anti-Inflammatory Diet (GrAID) — Specially designed diet based on the most recent scientific evidence of the inflammatory characteristics of food and food groups. Basically, subjects will be instructed to increase uptake of food components that hold potential anti-inflammatory proportions and to avoid food components that may showcase potential pro-inflammatory proportions.
  Arms: Groningen Anti-Inflammatory Diet (GrAID)
Dietary Supplement: ColoVit capsule — Vitamin B2/B3/C supplement in a ColoPulse-coated capsule
  Arms: ColoVit capsule
Other: ColoPulse-placebo capsule — A capsule containing microcrystalline cellulose which is coated using the same ColoPulse technology as is used with the ColoVit
  Arms: Placebo capsule

SUMMARY:
This study will evaluate if the Groningen Anti-Inflammatory Diet and the ileocolonic delivery of vitamin B2, B3 and C can positively influence the course of Crohn's disease and can positively alter the gut microbiome of Crohn's disease patients as well as healthy volunteers.

DETAILED DESCRIPTION:
It is becoming increasingly more well known that diet and the microbiome have a pivotal role in the development and course of inflammatory bowel diseases (IBD). Strict exclusive enteral nutrition (EEN) can induce remission in Crohn's Disease (CD) and is the standard treatment in paediatric CD. Implementing a restrictive diet in adults is difficult; adult patients do not tend to adhere to EEN. Recently, the CD-exclusion diet (CDED) combined with partial enteral nutrition demonstrated to be effective in CD-patients with flares.

Additionally, accumulating evidence suggests that intake of vitamins can influence disease course, mainly by beneficially modulating the gut microbiota and gut redox potential, especially if the vitamins can be delivered to the colon.

Nevertheless, no dietary guidelines are available to physicians and patients. Due to complaints of certain foods and patients' eagerness to postpone new flares, patients start experimenting with their food. As patients with CD are already often malnourished, this poorly substantiated experimenting puts them even more at risk for malnutrition and could have a potential negative effect on their disease outcomes. Next, quality of life of patients decreases and healthcare costs will rise. Therefore, both patients and physicians are in desperate need of evidence for an anti-inflammatory dietary advice in CD. As compliance to a diet increases when they are supported by family members, their household members will also be asked to participate in the study. Simultaneously studying their healthy family members will also provide information of the effect of this anti-inflammatory diet or intake of lieocolonic-delivered vitamins on their microbiome and markers of inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria CD patients:

* Participant understands the study procedures and signed an informed consent to participate in this study
* Previously diagnosed with CD; Montreal classification: L1 (Ileal), L2 (colonic), or L3 (ileocolonic).
* Low-mild disease activity (no clinically relevant symptoms and HBI<8 or CDAI <220)
* Evidence of mucosal inflammation (faecal calprotectin ≥100 μg/g)
* Able to attend to the outpatient clinic of the UMCG, Martini Hospital, MCL Leeuwarden or Isala
* ≥18 years of age
* Able to use oral feeding and willing to undergo a dietary intervention (Follow a diet or use a vitamin B2/B3/C supplement or placebo)

Inclusion Criteria healthy volunteers:

* Participant understands the study procedures and signed an informed consent to participate in this study
* Never been diagnosed with IBD or any other chronic inflammatory condition.
* Participant has no health conditions that would prevent him/her from fulfilling the study requirements as judged by the investigator on the basis of medical history and routine laboratory test results.
* Able to attend to the outpatient clinic of the UMCG, Martini Hospital, MCL Leeuwarden or Isala
* ≥18 year of age
* Able to use oral feeding and willing to undergo a dietary intervention (Follow a diet or use a vitamin B2/B3/C supplement or placebo)

Exclusion Criteria CD patients:

* Life expectancy <12 months
* Active Crohn's disease (HBI≥8 or CDAI>220), or expecting drug intervention within 3 months
* Colonoscopy and colon cleansing in the past 3 months;
* Use antibiotics, probiotics (eg Yakult, Vifit, Activia) or specific prebiotics supplements 3 weeks prior to the start of the intervention
* Use of vitamin/mineral supplements 1 week prior to the start of the intervention (except for vitamin D and/or calcium)
* Use Methotrexate drugs or chronic use of antacids, H2 or proton-pump inhibitors
* With a history of GI disorders or GI surgery that are likely to interfere with the pH-dependent mode of action of the Colovit-capsule
* Patients with a pouch or stoma
* Pregnant or breastfeeding (or foreseen pregnancy during dietary intervention period)
* Swallowing disorders, not able to tolerate oral food, or use of tube feeding (EEN)
* Previously proven anaphylactic reaction to foods included in the food boxes
* Previously diagnosed with Celiac Disease or following a gluten-free diet
* Following a vegetarian or vegan diet

Exclusion Criteria healthy subjects:

* Life expectancy <12 months
* Previously diagnosed with IBD or any other chronic inflammatory condition
* Colonoscopy and colon cleansing in the past 3 months;
* Use antibiotics, probiotics (eg Yakult, Vifit, Activia) or specific prebiotics supplements 3 weeks prior to the start of the intervention
* Use of vitamin/mineral supplements 1 week prior to the start of the intervention (except for vitamin D and/or calcium)
* With a history of GI disorders or taken drugs that are likely to interfere with mode of action of interventions, such as chronic use of antacids or proton-pump inhibitors
* Abnormal clinical chemistry and haematology laboratory test results of clinical significance that in the judgment of the investigator would interfere with the participant's ability to comply with the study protocol (which might confound the interpretation of the study results), or put the participant at undue risk.
* Presence of a stoma
* History or presence of cancer in the prior two years, except for non-melanoma skin cancer.
* Recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >60g (men) / 40g (women) pure alcohol per day (1.5 l / 1 l beer resp. 0.75 l / 0.5 l wine).
* Pregnant or breastfeeding (or foreseen pregnancy during dietary intervention period) The method of contraception must be recorded in the source documentation.
* Swallowing disorders, not able to tolerate oral food, or use of tube feeding (EEN)
* Previously proven anaphylactic reaction to foods included in the food boxes
* Previously diagnosed with Celiac Disease or following a gluten-free diet
* Following a vegetarian or vegan diet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in faecal calprotectin | Faeces sample collection at 4 time points: At baseline (0 months), after 3 months, after 6 months, after 12 months
  Primary outcome for CD patients
Change in microbiome composition measured by metagenomic sequencing- based profiles | Faeces sample collection at 3 time points: At baseline (0 months), after 3 months, after 12 months
  Primary outcome for healthy volunteers and CD patients

SECONDARY OUTCOMES:
The number of flares (defined as faecal calprotectin >200 μg/g and Crohn's Disease Activity Index (CDAI) ≥220 points) | Faeces sample collection and CDAI score determination at 4 time points: At baseline (0 months), after 3 months, after 6 months, after 12 months
  Secondary outcome for CD patients
Improvements of Quality of life scores as assessed by Inflammatory Bowel Disease Questionnaire (Score range of 32-224, The higher the score the higher the Quality of Life) | Questionnaires at 3 time points: At baseline (0 months), after 3 months, after 12 months
  Secondary outcome for CD patients
Improvements of Quality of life scores as assessed Food Related Quality of Life Questionnaire (Score range of 29-145, The higher the score the higher the Food related-Quality of Life) | Questionnaires at 3 time points: At baseline (0 months), after 3 months, after 12 months
  Secondary outcome for CD patients and healthy volunteers
Adherence to the dietary interventions as assessed by a Dietary Compliance Questionnaire | Questionnaires at 3 time points: At baseline (0 months), after 3 months, after 12 months
  Secondary outcome for CD patients and healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers outside of the study team.

REFERENCES:
- [Derived] Otten AT, Peters V, Barth I, Stevens CL, Bourgonje AR, Frijlink HW, Harmsen HJM, Rehman A, Campmans-Kuijpers MJE, Dijkstra G. Effects of ileocolonic delivered vitamin B2, B3 and C (ColoVit) or the Groningen anti-inflammatory diet on disease course and microbiome of patients with Crohn's disease (VITA-GrAID study): a protocol for a randomised and partially blinded trial. BMJ Open. 2023 Mar 14;13(3):e069654. doi: 10.1136/bmjopen-2022-069654. PMID 36918234